CLINICAL TRIAL: NCT06124963
Title: A Phase II Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of WX390 Combined With Toripalimab in Patients With Advanced Gastric-type Endocervical Adenocarcinoma With STK11 Mutations
Brief Title: A Study of WX390 Combined With Toripalimab in Patients With Advanced Gastric-type Endocervical Adenocarcinoma With STK11 Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JYP0390M207
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Gastric Type Adenocarcinoma (GAS) With STK11 Mutation
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: WX390 continuous oral dosing (0.9 mg once a day) Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX390 + Toripalimab (Experimental): Participants will receive WX390 continuous oral dosing (0.9 mg once a day) and Toripalimab fixed dose (240 mg, intravenous, Day 1, every 3 weeks).
  Interventions: Drug: WX390; Drug: Toripalimab

INTERVENTIONS:
Drug: WX390 — WX390 tablet, 0.9 mg once a day
  Other Names: WXFL10030390
Drug: Toripalimab — 240 mg, Day 1, every 3 weeks

SUMMARY:
The goal of this clinical trial is to evaluate the safety and preliminary efficacy of WX390 combined with Toripalimab in patients with advanced Gastric-type Endocervical Adenocarcinoma with STK11 mutations. The main questions it aims to answer are:

* Pharmacokinetic (PK) characteristics of WX390 combined with Toripalimab treatment.
* Safety and preliminary in combined therapy. Participants will be treated with WX390 orally and Toripalimab intravenously, and follow the efficacy and safety evaluation according to the protocol.

DETAILED DESCRIPTION:
This study will be an open-label, multicenter phase II clinical trial. After being informed about the study and potential risks, all patients giving written informed consent will undergo a 28-days screening period to determine eligibility for study entry. And then patents will be administered for 8 cycles treatment and 8 weeks safety follow up after the last dose of treatment. The efficacy and safety measures will be conducted and collected every cycle.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histological or cytological confirmed advanced Gastric-type Endocervical Adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of more than 3 months
* At least one measurable lesion according to RECIST 1.1
* Adequate organic function
* Signed and dated informed consent

Exclusion Criteria:

* Anti-cancer therapy within 30 days prior to the initiation of investigational treatment
* Major surgery within 30 days prior to the initiation of study treatment
* Received corticosteroids treatment or other immunodepressant within 2 weeks before the first dose of study treatment
* Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for alopecia)
* Patients who are suffering active interstitial lung disease
* Evidence of ongoing or active serious infection
* History of human immunodeficiency virus (HIV) infection or active hepatitis B or C infection
* Inability to take medication orally
* Abuse of alcohol or drugs
* People with cognitive and psychological abnormality or with low compliance
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate (PFS rate) | up to 24 weeks
  PFS rate, defined as the proportion of patients who have not experienced disease progression (PD) or death due to any cause during the study period.
Objective response rate (ORR) | up to 24 weeks
  ORR, defined as the percentage of participants with complete response (CR) or partial response (PR) confirmed by RECIST v1.1 assessment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 weeks
  PFS, defined as the time from the first treatment to the first occurrence of disease progression or death due to any cause during the study period (whichever comes first).
Overall survival (OS) | up to 48 weeks
  OS, defined as the time from the first treatment to death due to any cause.
Time to reach plasma Cmax (Tmax) of WX390 | up to 24 weeks
  Test the plasma drug concentration of WX390 to calculate Tmax.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kang, PhD, Principal Investigator — The Obstetrics & Gynecology Hospital of Fudan University (Shanghai Red House Ob & Gyn Hospital)
Locations (1):
- The Obstetrics & Gynecology Hospital of Fudan University (Shanghai Red House Ob & Gyn Hospital), Shanghai, Shanghai Municipality, China